CLINICAL TRIAL: NCT06911528
Title: A Prospective Study to Evaluate the Application of EndoScell Intraoperative Cellular Probing Technology in Breast Conserving Therapy and Sentinel Lymph Node Biopsy for Early-Stage Breast Cancer
Brief Title: Application of EndoScell Intraoperative Cellular Probing Technology for Early-Stage Breast Cancer
Acronym: EDGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jiong Wu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EDGE; HYXH2024012 (Other Grant/Funding Number: Shanghai Anticancer Development Foundation)
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer; Sentinel Lymph Node; Frozen Section; Cytology
Keywords: Breast carcinoma; sentinel lymph node; tracer; touch imprint cytology; epifluorescence widefield microscope system
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intraoperative Assessment (Experimental): After screening and enrollment, the EndoScell Scaner (ES) novel intraoperative cellular probing technology will be used for intraoperative evaluation of the sentinel lymph node. Concurrently, imprint cytology will be performed for evaluation. During the study period, intraoperative decisions will primarily reference the results of the imprint cytology technique.
  Interventions: Procedure: EndoScell Scaner (ES) novel intraoperative cellular probing technology

INTERVENTIONS:
Procedure: EndoScell Scaner (ES) novel intraoperative cellular probing technology — In this project, we utilize the miniature wide-angle focusing microscope for intraoperative cell-level observation and detection, a technology in which our hospital has conducted extensive research and accumulated rich experience.

SUMMARY:
Sentinel Lymph Node Biopsy (SLNB) is a common surgical treatment for breast cancer and a primary method for assessing the pathological status of axillary lymph nodes. Precise intraoperative detection of sentinel lymph nodes during surgery assists in timely evaluation of axillary lymph node pathology and helps in formulating further treatment strategies.

Touch imprint cytology (TIC) is one of the most commonly used intraoperative detection techniques. The new intraoperative cellular detection technology, EndoScell Scanner (ES), uses an improved real-time miniaturized fluorescence microscopy system for image acquisition. The ultra-high-resolution images obtained can reach the cellular level. In previous studies, the accuracy and sensitivity of this technology for intraoperative detection of sentinel lymph nodes were comparable to imprint cytology, but it is much more rapid. The detection technology uses fluorescein sodium and methylene blue as fluorescent dyes, which is non-invasive and also non-consumptive of tissue samples.

This study involves patients scheduled for sentinel lymph node biopsy and aims to evaluate the clinical application value of the EndoScell Scanner (ES) for intraoperative assessment of the pathological status of sentinel lymph nodes through a prospective self-controlled study. To avoid the potential impact of methylene blue on the ES detection technology, we will use mitoxantrone as a new dye for sentinel lymph node tracing in this study.

The primary study objective is to compare the accuracy of the ES detection technology in assessing sentinel lymph node status, using paraffin pathology examination as the gold standard. The primary endpoint is the accuracy of the ES technology. Secondary endpoints include the image quality score of the ES detection, the learning curve of the surgeons, and the time required for detection.

DETAILED DESCRIPTION:
In recent years, the incidence of breast cancer in China has risen rapidly. Over the past two decades, the annual average incidence rate has increased from 15 per 100,000 to about 30 per 100,000. In first-tier cities like Shanghai, the incidence rate even exceeds 60 per 100,000, making breast cancer the leading malignant tumor threatening women's health. Compared to Western countries, the onset age of breast cancer in Chinese women is relatively younger, with over 54% of cases occurring before menopause. Surgery remains the mainstay of comprehensive treatment for breast cancer. Nearly half of the patients require mastectomy due to the extent or location of the tumor, resulting in significant disfigurement and long-term psychological trauma. In recent years, the demand for postoperative breast appearance among breast cancer patients in China has been increasing, leading to a rise in the proportion of conventional breast-conserving surgery, breast-conserving surgery, and various types of breast reconstruction surgeries.

Breast-conserving surgery combined with postoperative radiotherapy can improve the postoperative breast appearance and quality of life while achieving tumor safety equal to or even better than that of total mastectomy. Breast-conserving oncoplastic surgery, which combine the principles of conventional breast conservation with plastic surgery techniques, further enhance the feasibility and safety of breast-conserving surgery.

The development of breast-conserving oncoplastic surgery has created a more urgent need to ensure negative margins intraoperatively. Despite expanding surgical indications due to the application of oncoplastic techniques, the positive margin rate of breast-conserving oncoplastic surgery is not significantly different from that of conventional breast-conserving surgery, ranging from 5% to 15%. Although re-excision after a positive margin does not affect local recurrence risk, it significantly diminishes postoperative cosmetic outcomes. More importantly, the design of oncoplastic surgery incisions becomes a challenge if mastectomy is needed based on margin status. Currently, the most accurate method for margin assessment is postoperative margin staining followed by radial sectioning and paraffin pathology examination. To enable timely intraoperative margin assessment, various methods have been proposed, including intraoperative frozen section analysis, specimen X-ray photography, and micro-computed tomography. However, these methods require ex vivo specimen evaluation and have limited sensitivity. Small sample studies have used micro-PET/CT technology for specimen imaging, but its high cost prevents widespread clinical validation and application.

The EndoScell Scaner (ES) is a novel intraoperative cell detection technology that uses a modified real-time miniaturized fluorescence microscope system for image acquisition, achieving ultra-high resolution at the cellular level. Previous studies have shown that its accuracy and sensitivity in intraoperative sentinel lymph node detection are comparable to those of cytological imprinting but with greater speed. This technology employs sodium fluorescein and methylene blue as fluorescent dyes, is non-invasive, and does not consume tissue samples.

This study aims to evaluate the clinical value of the EndoScell Scaner (ES) novel intraoperative cell probing technology for intraoperative margin assessment in patients undergoing conventional breast-conserving surgery and breast-conserving oncoplastic surgery combined with sentinel lymph node biopsy. The primary objective is to compare the accuracy of ES technology in assessing margin status and sentinel lymph node status using paraffin pathology as the gold standard. The primary endpoints are the accuracy of ES technology, positive margin rate, and reoperation rate; the secondary endpoints are ES detection image quality score, learning curve of surgeons, and detection time.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older (inclusive)
* Female
* Preoperative pathology confirmed invasive breast carcinoma or ductal carcinoma in situ
* Scheduled for sentinel lymph node biopsy
* Capable of and willing to provide informed consent

Exclusion Criteria:

* Patients with a confirmed allergy to methylene blue or sodium citrate tracers
* Pregnant or lactating women
* Patients unwilling to participate in the clinical study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 709 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy of ES technology | After the final pathological results are obtained, it is usually about 2 weeks after surgery
  the accuracy of the ES technology （including accuracy, sensitivity and specificity）
The reoperation rate | 3 months after surgery
  The proportion of reoperations due to a positive margin

SECONDARY OUTCOMES:
The quality score of ES imaging | After the final pathological results are obtained, it is usually about 2 weeks after surgery
  The image quality of ES was scored by the pathologist
The learning curve of the surgeons | through study completion, an average of 1 year
  Evaluate the number of cases required for the surgeon to achieve 95% or more accuracy
The time required for the intraoperative evaluation | through study completion, an average of 1 year
  The time required for intraoperative detection using ES technology

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol